CLINICAL TRIAL: NCT01458314
Title: Evaluation of the Additional Effect of Non Invasive Mechanical Ventilation During a Rehabilitative Program With Cycloergometer in Patients With Chronic Respiratory Insufficiency Using Nocturnal Home Ventilation
Brief Title: Non Invasive Mechanical Ventilation in Chronic Respiratory Insufficiency Patients During Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Salvatore Maugeri (Other)
Collaborators: Azienda Ospedaliero, Universitaria Pisana (Other); Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Michele Vitacca, Principal investigator, Fondazione Salvatore Maugeri
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTS/10/01
Record Dates: First submitted 2011-10-12; First posted 2011-10-24 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Respiratory Insufficiency
Keywords: Physical exercise; Rehabilitation; NIV
MeSH Terms: conditions — Motor Activity | interventions — Methods; Rehabilitation; Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rehabilitation without NIV (Active Comparator): A usual rehabilitative training will be performed in patients using nocturnal NIV, without adoption of daily NIV
  Interventions: Other: Rehabilitation without NIV
- Daily NIV during rehabilitation (Experimental): Daily NIV will be adopted during the rehabilitation program in patients already using nocturnal NIV
  Interventions: Other: Daily NIV during rehabilitation

INTERVENTIONS:
Other: Daily NIV during rehabilitation — Addition of non invasive mechanical ventilation (NIV) during daily rehabilitation in patients using nocturnal NIV
  Other Names: Group 1; Intervention
  Arms: Daily NIV during rehabilitation
Other: Rehabilitation without NIV — Training in patients without NIV adoption
  Other Names: Group 2; No intervention
  Arms: Rehabilitation without NIV

SUMMARY:
Patients with Chronic Obstructive Pulmonary Disease (COPD) and chronic respiratory insufficiency (CRI) have severe dyspnoea during exercise at low load. Physiological studies performed in these patients during a unique session of training have shown a positive effect on exercise tolerance if non-invasive mechanical ventilation (NIV) was added during incremental effort test or endurance. Menadue and coworkers (2009) have shown in CRI patients with hypercapnia, secondary to COPD or cifoscoliosis, that combination of NIV during arm effort test improved ability to perform the exercise. Similar result was not reached using NIV during walking. Further studies have underlined a positive effect of the ventilation therapy during exercise within specific programs of pulmonary rehabilitation (Corner 2009). Moreover, the addition of NIV to an exercise training (ET) program in COPD patients may produce greater benefits in exercise tolerance and quality of life than exercise training alone (Garrod 2000).

A great improvement in health-related quality of life, functional status and gas exchange in COPD patients with chronic hypercapnic respiratory failure with nocturnal NIV compared with patients in pulmonary rehabilitation alone has been also shown by Duieverman (2008). However, in the same study Duieverman did not show any significant difference between groups in terms of tolerance to effort test.

Aim of the study is to evaluate if application of daily NIV during physical training may increase the benefits of rehabilitation in CRI patients with nocturnal NIV compared with patients with nocturnal NIV performing training under spontaneous breathing.

DETAILED DESCRIPTION:
INTERVENTION

Group 1 (NIV during training + nocturnal NIV): This group of patients will use the usual NIV during night and will perform a rehabilitative program of at least 20 sessions of training at cycloergometer under NIV.

NO INTERVENTION

Group 2 (training in Spontaneous Breathing [SB] + nocturnal NIV): This group of patients will use the usual NIV during night and will be trained in a rehabilitative daily program without NIV. This group will be considered the "control" group.

Sessions: 30 minutes/session, 2 times/day, 4-5 times a week for a total of 20-25 session in 3 weeks.

Intensity: each patient will start at 50% of each individual's maximum work capacity (cycloergometer) increasing up to the maximum tolerated, according to Maltais's protocol.

NIV SETTING:

Training: Facial mask with usual setting (Inspiratory Positive Airway Pressure [IPAP] 10-15; Expiratory Positive Airway Pressure [EPAP] 4-6 cmH20) with a possible adjustment in agreement with the comfort.

The adjustment of ventilation during training will be only within the first 3 sessions according to the following protocol:

COPD patients: increase up to 3 cmH2Os of EPAP and decrease up to 3 cmH2Os of IPAP.

Restricted patients: increase up to 3 cmH2Os of IPAP.

Nocturnal ventilation: mask and usual setting

The primary outcome of the study is evaluation of effort tolerance measured by 6 minutes Walking Test (6-min Walking Test). The hypothesis is to verify a percentage of variation between the two groups equal to 10% after the rehabilitative program. To get a study power of 80% and an alpha error <5% 25 patients for group had to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* A total of 50 patients aging 40-79 years will be enrolled ( 8 out of 50 will be from FSM in Lumezzane)
* Patients with chronic respiratory insufficiency (CRI) in treatment with nocturnal NIV from at least six months;
* Clinical stability (absence of disease re-exacerbations from at least 4 weeks before the study).

Exclusion Criteria:

* Cardiac diseases: unstable and/or exercise angina, congestive heart failure cardiac, uncontrolled cardiac arrhythmias, sinus tachycardia at rest (HR >120 bpm), hypertension at rest and/or during effort not adequately checked by therapy
* Orthopaedic and/or neuromuscular illnesses.

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-03; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Effort tolerance measured by 6-minutes Walking test | After 3 weeks
  Changes from baseline in 6-minutes Walking test

SECONDARY OUTCOMES:
Maximal Inspiratory Pressure/Maximal Expiratory Pressure | After 3 weeks
Quality of life MRF 28 | After 3 weeks
Gas analysis | After 3 weeks
Effort tolerance evaluated by 6-minutes walking test | After 3 weeks
  Changes in 6-minutes walking test evaluated at the end of the program
Endurance at cycloergometer test | After 3 weeks
Effort tolerance measured by 6-minutes Walking test | Follow up at 3 months after the end of the protocol
  Changes in 6-minutes Walking test evaluated 3 months after the end of the protocol

CONTACTS AND LOCATIONS:
Overall Officials: Michele Vitacca, MD, Principal Investigator — Fondazione Salvatore Maugeri
Locations (1):
- Fondazione Salvatore Maugeri, Lumezzane, Brescia, Italy

REFERENCES:
- [Derived] Vitacca M, Kaymaz D, Lanini B, Vagheggini G, Ergun P, Gigliotti F, Ambrosino N, Paneroni M. Non-invasive ventilation during cycle exercise training in patients with chronic respiratory failure on long-term ventilatory support: A randomized controlled trial. Respirology. 2018 Feb;23(2):182-189. doi: 10.1111/resp.13181. Epub 2017 Sep 22. PMID 28940820